CLINICAL TRIAL: NCT01674049
Title: Nutrient Timing Following Resistance Exercise in Young Overweight and Obese Young Men With a Family History of Diabetes
Brief Title: Nutrient Timing Following Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 081025
Record Dates: First submitted 2012-08-24; First posted 2012-08-28 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes
Keywords: nutrition; nutrient; timing; diabetes; family history; dairy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Nutritional Status; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise and Immediate Nutrition (Experimental): 40 min of circuit-style resistance exercise and 600g low-fat chocolate milk immediately after the exercise bout
  Interventions: Dietary Supplement: Immediate Nutrition; Other: Resistance Exercise
- Exercise and Nutrition 3 hours Post-Bout (Active Comparator): 40 min of circuit-style resistance exercise and 600g low-fat chocolate milk three hours after the exercise bout
  Interventions: Dietary Supplement: Nutrition 3 hours Post-Bout; Other: Resistance Exercise

INTERVENTIONS:
Dietary Supplement: Immediate Nutrition — Nutritional supplement consumed either immediately following a 40min resistance exercise bout
  Arms: Exercise and Immediate Nutrition
Dietary Supplement: Nutrition 3 hours Post-Bout — Nutritional supplement (600g low-fat chocolate milk) consumed three hours after the exercise bout
  Arms: Exercise and Nutrition 3 hours Post-Bout
Other: Resistance Exercise — A single 40 minute circuit-style bout of resistance exercise

SUMMARY:
The purpose of the proposed study is to examine the timing of post-exercise feeding on 15 hours post-exercise glycemic control and metabolic flexibility and in overweight and obese young men with a family history of type 2 diabetes.

Aim 1 - To determine the temporal effects of post-exercise feeding (i.e., immediate post-exercise vs. 3 hours post-exercise) on glycemic control, peripheral insulin sensitivity, and metabolic flexibility (as evaluated by sleep RQ) in this same group of participants. We hypothesize that a 3 hour delay in nutrient ingestion will promote significantly greater improvements in glucose tolerance, metabolic flexibility, and peripheral insulin sensitivity both immediately and several hours post-ingestion.

DETAILED DESCRIPTION:
The proposed study is cross-sectional and utilizes a within-subject design to study young men under two different nutrient timing protocols, which are randomly-ordered and spaced at least 2 weeks apart.

1. Participants will be screened for eligibility via phone or email and scheduled for an initial visit, in order to consent to the study and undergo some basic baseline evaluations. We will rely on participant self-report to verify absence of chronic disease or drug use.
2. After consenting to the study, fasting blood glucose, height, weight, and air displacement plethysmography (BodPod®) will be conducted in the Clinical Exercise Physiology Laboratory at The George Washington University, in Washington, DC. These measures may occur on the same day as consent or at another scheduled time.
3. After screening, consenting, and baseline assessments, participants will undergo 2 experimental conditions, which will be randomly-ordered and approximately 2 weeks apart. If possible, both of these experimental visits will be scheduled shortly after the consent form is signed.
4. A registered dietitian will instruct participants to eat a standardized (35 kcal∙kg body weight-1∙day-1) diet comprising 60% carbohydrate, 20% protein, and 20% fat for 3 days prior to both experimental sessions. This instruction will be administered after the BodPod® assessment is completed.
5. Participants will report to the USDA Laboratory chamber at 7:30 AM for the experimental sessions. Height, weight blood pressure and heart rate will be measured, then a fasting blood sample (5 cc) will be obtained for determination of basal glucose & insulin concentrations. A Hidalgo Ambulatory Monitoring Sensor Array Vest (Equivital I: Hidalgo Ltd., Cambridge UK) will be worn by all participants measured in the calorimeter for the entire 48 period. This device measures heart rate (HR), heat flux, core body temperature, posture and physical activity (PA) from a built-in accelerometer.
6. Then, the sensor portion of the CGMS then will be placed subcutaneously and the CGMS calibrated with whole blood using the Accu-Check Advantage (Roche Diagnostics, Indianapolis, IL) glucometer. Participants will then enter the whole room calorimeter (metabolic chamber) and complete a hunger scale. Hunger will be evaluated 10-20 minutes before the start of each meal and 2 hours after the resistance exercise bout. On the first day, participants eat a standard breakfast provided by the USDA kitchen at approximately 7:45-8:00AM.
7. Gutierrez or a research assistant will take obtain glucometer readings before and 60 minutes after each meal to calibrate the the CGMS. These evaluations will occur 4-6 times over the course of the day.
8. Standardized meals (lunch at 11:00AM and dinner at 7:00PM) will be provided for subjects by the USDA. Blood samples (5 cc each) will be collected prior to and 120 minutes after breakfast and lunch; and prior to and 30-, 60-, 90-, and 120-min following the start of the evening meal for the determination of post-meal responses in glucose & insulin. A trained phlebotomist with at least 50 successful IV catheter placements will place an IV catheter into the participant's median antecubital vein before the evening meal to facilitate multiple draws after the meal.
9. On the second day, subjects will awake in the calorimeter at approximately 7:00 AM and a fasting blood sample (5 cc) will be obtained for determination of basal concentrations of glucose & insulin.
10. At about 7:30 AM, subjects will eat a standardized breakfast to be consumed by 8:00 AM. Two hours after a standardized lunch meal, served at 11:00AM, participants will perform one of the following resistance exercise nutrient-timing protocols: immediate post-exercise nutrition at approximately 2:00 PM 3 hour post exercise nutrition at approximately 5:00 PM). All participants will undergo both experimental conditions at different testing sessions.

ELIGIBILITY:
Inclusion Criteria:

* BMI= 18-30
* Report at least one first degree relative with family history of type 2 diabetes - Healthy with no self-report of diagnosis of chronic disease

Exclusion Criteria:

* Self-report prior diagnosis of cardiovascular disease, pulmonary disease, adult asthma, dyspnea on exertion, current bronchitis, pneumonia, or tuberculosis, vascular disease, any intercurrent infection, hematologic/oncologic, any metastatic malignancy, anemia (hematocrit <35), thrombocytopenia, neutropenia, hematologic malignancy, bleeding dyscrasias, neurologic disorder, endocrine disorder, chronic renal diseases
* Any illegal drug use
* Coumadin, heparin, beta blocker, growth hormone supplementation, or illegal drug use
* Skeletal-muscular injury in the last 6 months (including severe sprains, broken bones, and tendon or ligament injuries)
* Alcohol use in excess of 2 drinks per day
* Smokers

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 48 hours
  Continuous Glucose Monitoring was used for about 48 hours, from the time the participants entered the chamber on the control day through their release two days later

SECONDARY OUTCOMES:
Serum insulin | 2 hours post supplement ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Jean L Gutierrez, PhD, Principal Investigator — The George Washington University
Locations (1):
- The George Washington University, Washington D.C., District of Columbia, United States